CLINICAL TRIAL: NCT04197219
Title: Pembrolizumab With Axitinib in Recurrent Endometrial Cancer With Deficient Mismatch Repair System Post PD1 Exposure: Phase II Trial
Brief Title: Pembrolizumab With Axitinib in Recurrent Endometrial Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI is leaving institution
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4819
Record Dates: First submitted 2019-10-16; First posted 2019-12-13 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Recurrent Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — pembrolizumab; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab & axitinib (Experimental): All participants enrolled will receive pembrolizumab as standard of care (SOC) combined with axitinib. Axitinib will be self-administered orally twice daily at 5 mg. On days when both drugs are administered, axitinib will be administered first, followed by pembrolizumab. Treatment will continue until disease progression or unacceptable grade 3/4 toxicities. For patients with a complete response to therapy, maintenance therapy with both drugs will be continued for 12 months.
  Interventions: Drug: Pembrolizumab; Drug: Axitinib

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg IV day 1 of each cycle every 21 days
Drug: Axitinib — 5 mg PO BID continuously

SUMMARY:
The main purpose of this study is to see if adding the experimental medication, axitinib, to usual treatment with pembrolizumab will work better than pembrolizumab alone. The study team will look at overall safety and side effects of the combination of axitinib and pembrolizumab to see how well it is tolerated. Researchers will also want to take some research blood samples to explore what effects the combination of treatment has on participants' cells and immune system and to see if there are things in participants' blood that can predict a response or resistance to the combined treatment.

DETAILED DESCRIPTION:
This is a Phase 2, open label study of pembrolizumab in combination with axitinib in adult women with recurrent endometrial cancer with deficient mismatch repair system. Twenty-six participants in total will be enrolled into the study. All participants enrolled will receive pembrolizumab as standard of care combined with axitinib.

Axitinib is approved by the Food and Drug Administration (FDA) for treatment in certain participants with advanced renal cell cancer but is considered investigational (experimental) in this study. However, it is not FDA approved for recurrent endometrial cancer. Axitinib is a type of drug called a tyrosine kinase inhibitor. It is thought to work by blocking tumor vasculature and decreasing the blood supply to the tumor. Also it has been shown to improve the function of immune cells within the tumor which may enable them to kill the tumor.

Pembrolizumab is an immunotherapy that is FDA approved to treat participants with recurrent endometrial cancer with deficient mismatch repair system (dMMR). dMMR means having genetic changes within the tumor that make it unstable and potentially able to benefit from immunotherapy. Pembrolizumab works by improving the function of the immune cells enabling them to kill cancer cells.

Axitinib given in combination with pembrolizumab has not been tested for endometrial cancer. In this study the combination of axitinib and pembrolizumab is experimental because it is not approved by the Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have recurrent endometrial cancer with deficient mismatch repair system. Mismatch repair deficiency is defined by 1. Immunohistochemistry with loss of expression of one of these proteins in tumor tissue as defined by standard of care: MLH1, MSH2, MSH6 and PMS2, 2. Microstaellite (MSI) unstable by PCR per standard of care, 3. MSI high by next generation sequencing using commercial platform specifically CARIS, TEMPUS or Foundation testing.
* Subjects must have histologically confirmed endometrioid, clear cell, high grade serous, undifferentiated carcinoma or mixed histology.
* Must have had prior therapy with a PD1 inhibitor, pembrolizumab.
* Up to 5 prior lines of therapy are allowed.
* Prior anti-angiogenesis therapy is not allowed. Bevacizumab if given with chemotherapy in primary or adjuvant setting is allowed if treatment-free interval exceeded 6 months.
* Subjects must have measurable disease based on RECIST 1.1 with at least one target lesion.
* Subjects must have an ECOG performance status of 0-1.
* Subjects must have normal organ and marrow function as defined below within 14 days of enrollment unless otherwise indicated:

  * Hemoglobin ≥ 9.0 g/dl (may have been transfused)
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelet count ≥ 100,000/mcL
  * Total bilirubin ≤ 1.5 x the upper limit of normal (ULN) range
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN orAST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver).
  * Estimated Creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)
  * TSH within normal institutional limits. If elevated, patient can be eligible if evaluated by an endocrine specialist, placed on replacement therapy and deemed eligible with no current or prior autoimmune disease.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* Negative serum or urine pregnancy test at screening for women of childbearing potential.
* Willing to use highly effective contraception throughout the study and for at least 30 days after last treatment administration if childbearing potential exists
* Availability of an archival FFPE tumor tissue block from primary diagnosis specimen, metastatic, or recurrent site. If an FFPE tissue block cannot be provided then 15 unstained slides (10 minimum) will be acceptable. Please refer to the laboratory manual for complete details.
* Urinary protein <2+ by urine dipstick. If dipstick is >2+, then 24-hour urinary protein <2 g per 24 hours is required.
* No evidence of uncontrolled hypertension as documented by 2 baseline blood pressure (BP) readings taken at least 1 hour apart whether same visit or different visits. The baseline systolic BP readings must be <140 mm Hg, and the baseline diastolic BP readings must be <90 mm Hg. The use of antihypertensive medications to control BP is allowed.

Exclusion Criteria:

* Patients with sarcoma or carcinosarcoma
* Mismatch repair proficient tumors
* Patients with primary platinum refractory cancer defined as progressing during or within 3 months of completing primary platinum therapy.
* Prior anti-cancer therapy within 3 weeks prior to study enrollment.
* Known symptomatic brain metastases requiring steroids. Patients with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study enrollment, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and are neurologically stable.
* Patients having received prior therapy with PD1 or PDL1 or CTLA4 inhibitors or other immunotherapeutic agents except pembrolizumab.
* Patients having received prior anti-VEGF therapy as explained above
* Bowel obstruction (with or without gastrostomy tube) or inability to take oral medications
* Patients with a prior or current bowel perforation or fistula
* Uncontrolled hypertension defined as 140/90 or greater despite medical management with multiple medications
* ECOG performance >1
* Active autoimmune disease that might deteriorate when receiving an immune-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
* Patients currently on immunosuppressive therapy except:

  * Intra-nasal, inhaled, topical or local steroid injections (e.g., intra-articular injection)
  * Steroids as premedication for hypersensitivity reaction (e.g., CT scan premedication)."
  * Systemic corticosteroids at physiologic doses not exceeding 10 mg/day of prednisone or equivalent
* Patients who are pregnant or breast feeding.
* Known history of testing positive for HIV or known acquired immunodeficiency syndrome.
* Known history of immune-mediated colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis.
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: breast cancer in situ, cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Prior organ transplantation including allogenic stem-cell transplantation.
* Active infection requiring intravenous systemic therapy.
* Known hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
* Vaccination within 4 weeks of the first dose of treatment and while on trials is prohibited except for administration of inactivated vaccines.
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5 Grade ≥ 3)"
* Persistent toxicity related to prior therapy (NCI CTCAE v. 5 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
* Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Gastrointestinal abnormalities including:

  * Inability to take oral medication;
  * Requirement for intravenous alimentation;
  * Treatment for active peptic ulcer disease in the past 6 months;
  * Active gastrointestinal bleeding, unrelated to cancer, as evidenced by clinically significant hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy;
  * Malabsorption syndromes.
* Requirement of anticoagulant therapy with oral vitamin K antagonists. Low-dose anticoagulants for maintenance of patency of central venous access device or prevention of deep venous thrombosis is allowed. Therapeutic use of low molecular weight heparin is allowed.
* Evidence of inadequate wound healing.
* Grade >3 hemorrhage within 4 weeks of patient enrollment.
* Evidence of tumor involvement of the myocardium or pericardium or tumor thrombus extending to the heart.
* Ongoing known cardiac dysrhythmias of NCI CTCAE Grade >2 or prolongation of the QTc interval to >500 msec.
* Current use or anticipated need for treatment with drugs or foods that are known strong CYP3A4/5 inhibitors, including their administration within 10 days prior to patient enrollment (eg, grapefruit juice or grapefruit/grapefruit-related citrus fruits [eg, Seville oranges, pomelos], ketoconazole, miconazole, itraconazole, voriconazole, posaconazole, clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, amprenavir, fosamprenavir nefazodone, lopinavir, troleandomycin, mibefradil, and conivaptan). The topical use of these medications (if applicable), such as 2% ketoconazole cream, is allowed.
* Current use or anticipated need for drugs that are known strong CYP3A4/5 inducers, including their administration within 10 days prior to patient enrollment, eg, phenobarbital, rifampin, phenytoin, carbamazepine, rifabutin, rifapentin, clevidipine, St John's wort.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) at 12 weeks by RECIST 1.1 | Up to 12 weeks from start of treatment
  Percent of participants with ORR, defined as those having either a partial or complete response (according to RECIST 1.1) per investigator determination at 12 weeks from the date of study enrollment.
  Complete response (CR): Disappearance of all target lesions
  Partial response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD

SECONDARY OUTCOMES:
Average overall Survival (OS) | Assessed up to 60 months
  Average number in months from the date of study enrollment to the date of death (any cause) or last known date of follow up if otherwise lost to follow up.
Clinical benefit rate | Up to 12 weeks from start of treatment
  Clinical benefit, defined by percent of participants with ORR and stable disease at 12 weeks
Number of participants with grade 3 and 4 immune and non-immune related toxicities assessed via NCI CTCAE v.5.03 | 90 days from end of treatment
  Number of participants with grade 3 and 4 immune and non-immune related toxicities assessed via National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v.5.03
Average progression-free survival (PFS) | 12 months from end of treatment
  Average number of months from the date of study enrollment to the date of an event of disease progression (according to RECIST 1.1) per investigator determination or to the date of death (any cause).

OTHER OUTCOMES:
Translational endpoints | 12 months from end of treatment
  Translational markers to predict resistance and response to therapy. Identify genomic, immune related markers that can predict response and/or resistance to the combined therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Haider Mahdi, MD, Principal Investigator — Cleveland Clinic Women's Health Institute

IPD SHARING:
Plan to Share IPD: No
This is a single institution study and the IPD data are not planned to be shared outside the institution.

REFERENCES:
- [Background] Dellinger TH, Monk BJ. Systemic therapy for recurrent endometrial cancer: a review of North American trials. Expert Rev Anticancer Ther. 2009 Jul;9(7):905-16. doi: 10.1586/era.09.54. PMID 19589030
- [Background] Dizon DS. Treatment options for advanced endometrial carcinoma. Gynecol Oncol. 2010 May;117(2):373-81. doi: 10.1016/j.ygyno.2010.02.007. Epub 2010 Mar 12. PMID 20223510
- [Background] Bradford LS, Rauh-Hain JA, Schorge J, Birrer MJ, Dizon DS. Advances in the management of recurrent endometrial cancer. Am J Clin Oncol. 2015 Apr;38(2):206-12. doi: 10.1097/COC.0b013e31829a2974. PMID 23764681
- [Background] Alexandrov LB, Nik-Zainal S, Wedge DC, Aparicio SA, Behjati S, Biankin AV, Bignell GR, Bolli N, Borg A, Borresen-Dale AL, Boyault S, Burkhardt B, Butler AP, Caldas C, Davies HR, Desmedt C, Eils R, Eyfjord JE, Foekens JA, Greaves M, Hosoda F, Hutter B, Ilicic T, Imbeaud S, Imielinski M, Jager N, Jones DT, Jones D, Knappskog S, Kool M, Lakhani SR, Lopez-Otin C, Martin S, Munshi NC, Nakamura H, Northcott PA, Pajic M, Papaemmanuil E, Paradiso A, Pearson JV, Puente XS, Raine K, Ramakrishna M, Richardson AL, Richter J, Rosenstiel P, Schlesner M, Schumacher TN, Span PN, Teague JW, Totoki Y, Tutt AN, Valdes-Mas R, van Buuren MM, van 't Veer L, Vincent-Salomon A, Waddell N, Yates LR; Australian Pancreatic Cancer Genome Initiative; ICGC Breast Cancer Consortium; ICGC MMML-Seq Consortium; ICGC PedBrain; Zucman-Rossi J, Futreal PA, McDermott U, Lichter P, Meyerson M, Grimmond SM, Siebert R, Campo E, Shibata T, Pfister SM, Campbell PJ, Stratton MR. Signatures of mutational processes in human cancer. Nature. 2013 Aug 22;500(7463):415-21. doi: 10.1038/nature12477. Epub 2013 Aug 14. PMID 23945592
- [Background] Howitt BE, Shukla SA, Sholl LM, Ritterhouse LL, Watkins JC, Rodig S, Stover E, Strickland KC, D'Andrea AD, Wu CJ, Matulonis UA, Konstantinopoulos PA. Association of Polymerase e-Mutated and Microsatellite-Instable Endometrial Cancers With Neoantigen Load, Number of Tumor-Infiltrating Lymphocytes, and Expression of PD-1 and PD-L1. JAMA Oncol. 2015 Dec;1(9):1319-23. doi: 10.1001/jamaoncol.2015.2151. PMID 26181000
- [Background] Le DT, Durham JN, Smith KN, Wang H, Bartlett BR, Aulakh LK, Lu S, Kemberling H, Wilt C, Luber BS, Wong F, Azad NS, Rucki AA, Laheru D, Donehower R, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Greten TF, Duffy AG, Ciombor KK, Eyring AD, Lam BH, Joe A, Kang SP, Holdhoff M, Danilova L, Cope L, Meyer C, Zhou S, Goldberg RM, Armstrong DK, Bever KM, Fader AN, Taube J, Housseau F, Spetzler D, Xiao N, Pardoll DM, Papadopoulos N, Kinzler KW, Eshleman JR, Vogelstein B, Anders RA, Diaz LA Jr. Mismatch repair deficiency predicts response of solid tumors to PD-1 blockade. Science. 2017 Jul 28;357(6349):409-413. doi: 10.1126/science.aan6733. Epub 2017 Jun 8. PMID 28596308
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Background] Ott PA, Bang YJ, Berton-Rigaud D, Elez E, Pishvaian MJ, Rugo HS, Puzanov I, Mehnert JM, Aung KL, Lopez J, Carrigan M, Saraf S, Chen M, Soria JC. Safety and Antitumor Activity of Pembrolizumab in Advanced Programmed Death Ligand 1-Positive Endometrial Cancer: Results From the KEYNOTE-028 Study. J Clin Oncol. 2017 Aug 1;35(22):2535-2541. doi: 10.1200/JCO.2017.72.5952. Epub 2017 May 10. PMID 28489510
- [Background] United States Package Insert for Inlyta, dated January 2012
- [Background] Hutson TE, Lesovoy V, Al-Shukri S, Stus VP, Lipatov ON, Bair AH, Rosbrook B, Chen C, Kim S, Vogelzang NJ. Axitinib versus sorafenib as first-line therapy in patients with metastatic renal-cell carcinoma: a randomised open-label phase 3 trial. Lancet Oncol. 2013 Dec;14(13):1287-94. doi: 10.1016/S1470-2045(13)70465-0. Epub 2013 Oct 25. PMID 24206640
- [Background] Rini BI, Escudier B, Tomczak P, Kaprin A, Szczylik C, Hutson TE, Michaelson MD, Gorbunova VA, Gore ME, Rusakov IG, Negrier S, Ou YC, Castellano D, Lim HY, Uemura H, Tarazi J, Cella D, Chen C, Rosbrook B, Kim S, Motzer RJ. Comparative effectiveness of axitinib versus sorafenib in advanced renal cell carcinoma (AXIS): a randomised phase 3 trial. Lancet. 2011 Dec 3;378(9807):1931-9. doi: 10.1016/S0140-6736(11)61613-9. Epub 2011 Nov 4. PMID 22056247
- [Background] Inlyta Summary of Product Chracteristics, Pfizer Inc. http://www.ema.europa.eu/docs/en_GB/document_library/EPAR_-_Product_Informatio n/human/002406/WC500132188.pdf
- [Background] Aghajanian C, Sill MW, Darcy KM, Greer B, McMeekin DS, Rose PG, Rotmensch J, Barnes MN, Hanjani P, Leslie KK. Phase II trial of bevacizumab in recurrent or persistent endometrial cancer: a Gynecologic Oncology Group study. J Clin Oncol. 2011 Jun 1;29(16):2259-65. doi: 10.1200/JCO.2010.32.6397. Epub 2011 May 2. PMID 21537039
- [Background] Bender D, Sill MW, Lankes HA, Reyes HD, Darus CJ, Delmore JE, Rotmensch J, Gray HJ, Mannel RS, Schilder JM, Hunter MI, McCourt CK, Samuelson MI, Leslie KK. A phase II evaluation of cediranib in the treatment of recurrent or persistent endometrial cancer: An NRG Oncology/Gynecologic Oncology Group study. Gynecol Oncol. 2015 Sep;138(3):507-12. doi: 10.1016/j.ygyno.2015.07.018. Epub 2015 Jul 15. PMID 26186911
- [Background] Wong C, Wellman TL, Lounsbury KM. VEGF and HIF-1alpha expression are increased in advanced stages of epithelial ovarian cancer. Gynecol Oncol. 2003 Dec;91(3):513-7. doi: 10.1016/j.ygyno.2003.08.022. PMID 14675669
- [Background] Yamamoto S, Konishi I, Mandai M, Kuroda H, Komatsu T, Nanbu K, Sakahara H, Mori T. Expression of vascular endothelial growth factor (VEGF) in epithelial ovarian neoplasms: correlation with clinicopathology and patient survival, and analysis of serum VEGF levels. Br J Cancer. 1997;76(9):1221-7. doi: 10.1038/bjc.1997.537. PMID 9365173
- [Background] Brustmann H. Vascular endothelial growth factor expression in serous ovarian carcinoma: relationship with topoisomerase II alpha and prognosis. Gynecol Oncol. 2004 Oct;95(1):16-22. doi: 10.1016/j.ygyno.2004.07.040. PMID 15385105
- [Background] Manenti L, Paganoni P, Floriani I, Landoni F, Torri V, Buda A, Taraboletti G, Labianca R, Belotti D, Giavazzi R. Expression levels of vascular endothelial growth factor, matrix metalloproteinases 2 and 9 and tissue inhibitor of metalloproteinases 1 and 2 in the plasma of patients with ovarian carcinoma. Eur J Cancer. 2003 Sep;39(13):1948-56. doi: 10.1016/s0959-8049(03)00427-1. PMID 12932675
- [Background] Kraft A, Weindel K, Ochs A, Marth C, Zmija J, Schumacher P, Unger C, Marme D, Gastl G. Vascular endothelial growth factor in the sera and effusions of patients with malignant and nonmalignant disease. Cancer. 1999 Jan 1;85(1):178-87. PMID 9921991
- [Background] Mesiano S, Ferrara N, Jaffe RB. Role of vascular endothelial growth factor in ovarian cancer: inhibition of ascites formation by immunoneutralization. Am J Pathol. 1998 Oct;153(4):1249-56. doi: 10.1016/S0002-9440(10)65669-6. PMID 9777956
- [Background] Ohm JE, Carbone DP. VEGF as a mediator of tumor-associated immunodeficiency. Immunol Res. 2001;23(2-3):263-72. doi: 10.1385/IR:23:2-3:263. PMID 11444391
- [Background] Gabrilovich D, Ishida T, Oyama T, Ran S, Kravtsov V, Nadaf S, Carbone DP. Vascular endothelial growth factor inhibits the development of dendritic cells and dramatically affects the differentiation of multiple hematopoietic lineages in vivo. Blood. 1998 Dec 1;92(11):4150-66. PMID 9834220
- [Background] Terme M, Pernot S, Marcheteau E, Sandoval F, Benhamouda N, Colussi O, Dubreuil O, Carpentier AF, Tartour E, Taieb J. VEGFA-VEGFR pathway blockade inhibits tumor-induced regulatory T-cell proliferation in colorectal cancer. Cancer Res. 2013 Jan 15;73(2):539-49. doi: 10.1158/0008-5472.CAN-12-2325. Epub 2012 Oct 29. PMID 23108136
- [Background] Ohm JE, Gabrilovich DI, Sempowski GD, Kisseleva E, Parman KS, Nadaf S, Carbone DP. VEGF inhibits T-cell development and may contribute to tumor-induced immune suppression. Blood. 2003 Jun 15;101(12):4878-86. doi: 10.1182/blood-2002-07-1956. Epub 2003 Feb 13. PMID 12586633
- [Background] Bouzin C, Brouet A, De Vriese J, Dewever J, Feron O. Effects of vascular endothelial growth factor on the lymphocyte-endothelium interactions: identification of caveolin-1 and nitric oxide as control points of endothelial cell anergy. J Immunol. 2007 Feb 1;178(3):1505-11. doi: 10.4049/jimmunol.178.3.1505. PMID 17237399
- [Background] Ozao-Choy J, Ma G, Kao J, Wang GX, Meseck M, Sung M, Schwartz M, Divino CM, Pan PY, Chen SH. The novel role of tyrosine kinase inhibitor in the reversal of immune suppression and modulation of tumor microenvironment for immune-based cancer therapies. Cancer Res. 2009 Mar 15;69(6):2514-22. doi: 10.1158/0008-5472.CAN-08-4709. Epub 2009 Mar 10. PMID 19276342
- [Background] Kwilas AR, Ardiani A, Donahue RN, Aftab DT, Hodge JW. Dual effects of a targeted small-molecule inhibitor (cabozantinib) on immune-mediated killing of tumor cells and immune tumor microenvironment permissiveness when combined with a cancer vaccine. J Transl Med. 2014 Nov 13;12:294. doi: 10.1186/s12967-014-0294-y. PMID 25388653
- [Background] Kwilas AR, Donahue RN, Tsang KY, Hodge JW. Immune consequences of tyrosine kinase inhibitors that synergize with cancer immunotherapy. Cancer Cell Microenviron. 2015;2(1):e677. doi: 10.14800/ccm.677. PMID 26005708
- [Background] Laubli H, Muller P, D'Amico L, Buchi M, Kashyap AS, Zippelius A. The multi-receptor inhibitor axitinib reverses tumor-induced immunosuppression and potentiates treatment with immune-modulatory antibodies in preclinical murine models. Cancer Immunol Immunother. 2018 May;67(5):815-824. doi: 10.1007/s00262-018-2136-x. Epub 2018 Feb 27. PMID 29487979
- [Background] Bose A, Lowe DB, Rao A, Storkus WJ. Combined vaccine+axitinib therapy yields superior antitumor efficacy in a murine melanoma model. Melanoma Res. 2012 Jun;22(3):236-43. doi: 10.1097/CMR.0b013e3283538293. PMID 22504156
- [Background] Stehle F, Schulz K, Fahldieck C, Kalich J, Lichtenfels R, Riemann D, Seliger B. Reduced immunosuppressive properties of axitinib in comparison with other tyrosine kinase inhibitors. J Biol Chem. 2013 Jun 7;288(23):16334-16347. doi: 10.1074/jbc.M112.437962. Epub 2013 Apr 26. PMID 23625925
- [Background] Atkins MB, Plimack ER, Puzanov I, Fishman MN, McDermott DF, Cho DC, Vaishampayan U, George S, Olencki TE, Tarazi JC, Rosbrook B, Fernandez KC, Lechuga M, Choueiri TK. Axitinib in combination with pembrolizumab in patients with advanced renal cell cancer: a non-randomised, open-label, dose-finding, and dose-expansion phase 1b trial. Lancet Oncol. 2018 Mar;19(3):405-415. doi: 10.1016/S1470-2045(18)30081-0. Epub 2018 Feb 10. PMID 29439857
- [Background] Rini BI, Plimack ER, Stus V, Gafanov R, Hawkins R, Nosov D, Pouliot F, Alekseev B, Soulieres D, Melichar B, Vynnychenko I, Kryzhanivska A, Bondarenko I, Azevedo SJ, Borchiellini D, Szczylik C, Markus M, McDermott RS, Bedke J, Tartas S, Chang YH, Tamada S, Shou Q, Perini RF, Chen M, Atkins MB, Powles T; KEYNOTE-426 Investigators. Pembrolizumab plus Axitinib versus Sunitinib for Advanced Renal-Cell Carcinoma. N Engl J Med. 2019 Mar 21;380(12):1116-1127. doi: 10.1056/NEJMoa1816714. Epub 2019 Feb 16. PMID 30779529